CLINICAL TRIAL: NCT05563532
Title: The Effect of Maternal Dental Anxiety and Oral Hygiene Status on the Dental Anxiety and Periodontal Health of Their Children
Brief Title: Dental Anxiety and Periodontal Health
Status: Completed | Type: Observational
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Ekin Besiroglu, assistant profesor, Okan University
Other Study IDs: 2019/104.25
Record Dates: First submitted 2022-09-17; First posted 2022-10-03 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Dental Anxiety; Periodontal Health; Oral Hygiene
MeSH Terms: interventions — Oral Hygiene

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- anxious group: Children with a score ≥4 on the venham picture test were included.
  Interventions: Behavioral: dental anxiety and oral hygiene
- non-anxious group: Children with a score <4 on the venham picture test were included.

INTERVENTIONS:
Behavioral: dental anxiety and oral hygiene — Evaluation of the effect of mothers' dental anxiety and oral hygiene on children's dental anxiety and periodontal status.
  Groups: anxious group

SUMMARY:
Mothers usually have the primary role in bringing up children and developing health-related behaviors. The aim of this study was to determine the effect of mothers' dental anxiety and oral hygiene on the dental anxiety and periodontal health of their children.

The study included 280 randomly selected children, aged 4-12 years, who came to the dentist for the first time and their mothers. Demographic and oral hygiene information of the mothers was collected through a questionaire. Dental anxiety of the mothers and children was assessed using the Modified Dental Anxiety Scale (MDAS) and the Venham Picture Test (VPT), respectively.

DETAILED DESCRIPTION:
Anxiety is a neurotic syndrome in which patients have difficulty in explaining internal restlessness, anxiety and fear reaching the level of panic, which causes physiological and behavioral disorders as a result of affecting motor tension and even autonomic hyperactivity. Anxiety and fear are frequently encountered in dentistry clinical practice in both adults and children. Dental anxiety is also defined as intense fear and anxiety that occurs as a result of the thought that patients will be harmed, that they will have an unknown operation outside their control, and because they have had previous negative dental treatment experiences.

Direct factors such as previous traumatic dental experiences, postoperative complications, age, gender, anxious temperament in childhood, and indirect factors such as the effect of family on the approach to dental treatment and sociodemographic factors have been reported to have an effect on the development of dental anxiety. Most early school-age children begin to imitate their parents as role models. Children in this age group internalize their mothers' values, attitudes and behaviors, since they usually spend more time with their mothers. It is thought that especially parents' dental anxiety may have an effect on their children's dental anxiety through modeling and knowledge.

Children with dental anxiety try every way to avoid dental treatment. The thought that patients will feel more pain than normal due to the anxiety they experience during dental treatments makes treatment difficult. Anxiety might lead to individuals discontinuing treatment, thereby worsening their dental health. As a result, necessary dental treatment becomes more time-consuming, invasive, and costly. At the same time, treatment anxiety impedes the clinical process, jeopardizes treatment results, and causes professional stress for dentists.

Dental anxiety is evaluated through projective tests, behavioral assessments, psychometric assessments, and physiological techniques. Behavioral assessment is based on the dentist or researchers scoring the behaviors visually. For this purpose, the Frankl Behavior Scale and the Yale Preoperative Anxiety Scale are used. Psychometric assessments are made with questionnaires, which are the most preferred because of their ease of application, and these are used to measure the anxiety of children or adults before dental treatment. At the present time, the Modified Dental Anxiety Scale (MDAS) is frequently used for adults, while the Children's Fear Survey Schedule-Dental Subscale (CFSS-DS) is used for children. Projective techniques also use pictures or narratives of objects that may cause anxiety and fear in young children. The Venham Picture Test (VPT) and Children's Dental Fear Picture Test are commonly used projective techniques. Physiological techniques measure anxiety-related parameters such as salivary cortisol level, blood pressure, and dorsal skin response. However, it is thought that the equipment used in this technique may increase anxiety, especially in children.

From a review of literature it can be seen that there are few studies conducted in Turkey which have evaluated the effect of the mother on the child's dental anxiety and oral hygiene. The aim of this study was to determine the effects of mothers' dental anxiety and oral hygiene on the dental anxiety and periodontal health of their children, using psychometric analysis and projective methods.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for children were defined as age 4-12 years,
* Having no known systemic disease,
* visiting a dentist for the first time,
* not having reported acute pain.

Exclusion Criteria:

* The exclusion criteria for children were defined as having systemic disease,
* Having reported acute pain.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study inclusion criteria for mothers were the absence of any systemic and psychiatric disorders, not being pregnant or breastfeeding, non-smoking, not having received periodontal treatment in the last 6 months, and with at least 20 teeth and willing to participate in the study. The inclusion criteria for children were defined as age 4-12 years, having no known systemic disease, visiting a dentist for the first time, and not having reported acute pain. Only one child per family was included in the study for mother-child pairs.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of the child's dental anxiety level | 2 years
  The Venham Picture Test (VPT) was applied to the children to determine dental anxiety levels. The VPT consists of eight illustrations of human figures expressing various emotional reactions. The child selects pictures to reflect their current emotions. Each picture of an anxious child is assigned a score of 1, and each picture of a non-anxious child is assigned a score of 0. The total score ranges from 0 to 8, with a high score indicating a high level of anxiety, and a score of ≥4 is evaluated as high level dental anxiety. The children were separated into two groups based on whether or not they were classified as anxious.

SECONDARY OUTCOMES:
Evaluation of the mother's dental anxiety level | 2 years
  Modified Dental Anxiety Scale (MDAS) was applied to the mothers to determine dental anxiety levels. The MDAS consists of 5 items providing a total score ranging from 5 to 25 points. A MDAS score ≥19 is evaluated as a high level of dental anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Okan university, Istanbul, Tuzla, Turkey (Türkiye)

REFERENCES:
- [Derived] Besiroglu-Turgut E, Kayaalti-Yuksek S, Bulut M. Evaluation of the relationship between dental anxiety and oral health status of mothers and their children. BMC Oral Health. 2024 Jun 28;24(1):749. doi: 10.1186/s12903-024-04530-0. PMID 38943136